CLINICAL TRIAL: NCT04761536
Title: Volume-outcome Relationship in Rectal Cancer Surgery
Status: Completed | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Giuseppe Sigismondo Sica, MD, PhD, Associate Professor, University of Rome Tor Vergata
Other Study IDs: REGISTROSPERIMENTAZIONI XX/21
Record Dates: First submitted 2021-02-15; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Rectal Cancer; Anastomotic Leak Rectum
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: patients undergoing ARR with primary anastomosis between November 2016 and December 2020 after centralization of rectal cancer cases
  Interventions: Other: Rectal cancer case centralization
- B: patients undergoing ARR with primary anastomosis between January 2006 and October 2016

INTERVENTIONS:
Other: Rectal cancer case centralization — In November 2016, the decision to centralize rectal cancer patients to only one surgical unit was taken, with only two surgeons performing the procedures. Furthermore, a close collaboration with local Gastroenterology Units and General Practiotioners was started in order to increase colorectal cancer case referral to our unit. At the same time, we decided to promote the use of laparoscopy and to implement ERAS protocol in our colorectal surgery practice.
  Groups: A

SUMMARY:
Hospital centralization effect is reported to lower complications and mortality especially for high risk and complex general surgery operations, including colorectal surgery. However, no linear relation between volume and outcome has been demonstrated. Aim of the study was to evaluate the increased surgical volume effect on early outcomes of patient undergoing restorative anterior rectal resection (ARR).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of a cancer located in the rectum, defined according to the international definition by D'Souza et al.,
* elective setting
* anterior rectal resection with primary anastomosis (with or without diverting loop ileostomy).

Exclusion Criteria:

* age below age of 18,
* inflammatory bowel disease,
* acquired or congenital immunodeficiency,
* preoperative infection,
* pregnancy,
* ASA IV,
* presence of synchronous cancers,
* abdominoperineal resection (APR),
* failure to perform rectal resection and primary anastomosis,
* emergency setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study involved all consecutive eligible patients undergoing elective restorative anterior rectal resection (ARR) for rectal cancer between November 2016 and December 2020 in our Minimally Invasive Surgery Unit of Tor Vergata University Hospital unit (Group A). Outcomes for Group A were compared with an historical control group, consisting of all consecutive patients undergoing ARR in the same hospital between January 2006 and October 2016 (Group B).
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Anastomotic leak | up to 30 days after discharge
  rate of any postoperative leakage of colo-rectal anastomosis clinically, radiologically or endoscopically demonstrated

SECONDARY OUTCOMES:
Postoperative complications | up to 30 days after discharge
  rate of any surgical site infection clinically demonstrated
Surgical site infection | up to 30 days after discharge
  Rate of any complication after rectal resection
Pneumonia | up to 30 days after discharge
  rate of radiologically demonstrated pneumonia
Ileus | up to 30 days after discharge
  rate of any ileus clinically demonstrated
Bleeding | up to 30 days after discharge
  Rate of any clinically radiologically or endoscopically demonstrated bleeding after rectal resection
Reoperation | up to 30 days after discharge
  Rate of any reoperation
Readmission | up to 90 days after discharge
  Rate of any unplanned readmission after discharge
30-days-mortality | up to 30 days after discharge
  Rate of any mortality
1-year stoma persistence | up to one year after surgery
  rate of stoma persistence
Length of hospital stay | up to 30 days after discharge
  number of days between primary rectal resection and discharge
Use of minimally invasive approach | up to 30 days after discharge
  rate of minimally invasive rectal ARR performed
Operative time | up to 30 days after discharge
  Mean operative time
Conversion to open surgery | up to 30 days after discharge
  rate of conversion form laparoscopy to one surgery
need of postoperative blood transfusion | up to 30 days after discharge
  rate of postoperative transfusion